CLINICAL TRIAL: NCT06079788
Title: Study of Adrenocorticotropic Hormone on Children With Frequent Relapse or Steroid-dependent Nephrotic Syndrome: a Prospective, Multicenter, Randomized，Open-label Clinical Trial.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mao Jianhua (Other)
Collaborators: Tongji Hospital (Other); Children's Hospital affiliated to Capital Institute of Pediatrics (Unknown); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Children's Hospital of Nanjing Medical University (Other); Kunming Children's Hospital (Other); Yuying Childrens Hospital of Wenzhou Medical University (Unknown); Ningbo Women & Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Mao Jianhua, professor, The Children's Hospital of Zhejiang University School of Medicine
Organization: The Children's Hospital of Zhejiang University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAIR
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Nephrotic Syndrome in Children
Keywords: Nephrotic Syndrome; Frequently Relapsing Nephrotic Syndrome; Steroid Dependent Nephrotic Syndrome; Adrenocorticotropic Hormone
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Adrenocorticotropic Hormone; Steroids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adrenocorticotrophic Hormone Group (Experimental): ACTH 2 IU/kg/ day, qd,（the maximum dose ≤ 50 IU）, 28 days of continuous use for 5 days， for 24 weeks.
  Prednisone: 5mg；Oral tablets; 1.5-2 mg/kg, qod or 0.75-1mg/kg/day,qd
  Interventions: Drug: Adrenocorticotrophic Hormone
- Steroid Group (Active Comparator): Prednisone: 5mg；Oral tablets; 1.5-2 mg/kg, qod or 0.75-1mg/kg/day,qd, then gradually taper the steroid by 0.25mg/kg （qod） or 0.125mg/kg （qd） every 4 weeks.
  Interventions: Drug: Steroid

INTERVENTIONS:
Drug: Adrenocorticotrophic Hormone — For patients in complete remission, ACTH is given at a prednisone dose of 1.5-2mg/kg qod or 0.75-1mg/kg qd. ACTH 2 IU/kg/ day, qd,（the maximum dose ≤ 50 IU）, 28 days of continuous use for 5 days， for 24 weeks.
  Prednisone: 5mg；Oral tablets; 1.5-2 mg/kg, qod or 0.75-1mg/kg/day,qd, then gradually taper the steroid by 0.25mg/kg qod or 0.125mg/kg qd every 4 weeks.If stable, taper to 5mg qod (body surface area > 1.0m2) and 2.5mg qod (body surface area < 1.0m2) and maintain the dose until study completion.
  Other Names: ACTH
  Arms: Adrenocorticotrophic Hormone Group
Drug: Steroid — For patients in complete remission, Prednisone: 5mg；Oral tablets; 1.5-2 mg/kg, qod or 0.75-1mg/kg/day,qd, then gradually taper the steroid by 0.25mg/kg qod or 0.125mg/kg qd every 4 weeks. If stable, taper to 5mg qod (body surface area > 1.0m2) and 2.5mg qod (body surface area < 1.0m2) and maintain the dose until study completion.
  Arms: Steroid Group

SUMMARY:
Primary nephrotic syndrome accounts for approximately 90% of the total number of nephrotic syndrome in childhood and it is the most common glomerular disease in children. Although treatment with steroids is useful for primary nephrotic syndrome, proving to cause frequent relapse/steroid-dependent nephrotic syndrome after treatment and the usage of immunosuppressive agents has become a new choice for the treatment of such patients. This study is a prospective, multicenter, randomized，open-label clinical trial, evaluating the efficacy and safety of steroid combined with adrenocorticotrophic hormone（ACTH） to children who with frequently relapsing or steroid-dependent nephrotic syndrome, all we wish to obtain the proper drug choice and individualized treatment options for children with nephrotic syndrome.

DETAILED DESCRIPTION:
Although steroids are recognized as first-line treatments for nephrotic syndrome, the vast majority of children relapse, and about half of them have frequent relapse or steroids dependence after treatment with steroids alone. Some children experienced steroids-resistance after multiple relapses, and eventually developed into chronic kidney dysfunction. Long-term or repeated application of large doses of steroids will lead to side effects such as obesity, growth retardation, and hypertension. Although the treatment of steroids with immunosuppressive agents is a new choice for the treatment of such patients, traditional immunosuppressive agents will bring some serious irreversible side effects.

The clinical application of ACTH in children with nephrotic syndrome dates back to the late 1940s. In recent years, the new mechanism of action of ACTH is also being explored. A number of clinical studies on the treatment of nephrotic syndrome by ACTH have found that it can still achieve good efficacy in patients who are ineffective in first-line treatment. This study evaluated the efficacy of ACTH in the treatment of relapsing or steroid-dependent nephrotic syndrome in children, in order to provide a more effective and safer treatment for children with nephrotic syndrome as well as the therapeutic medication options.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2-14 years old;
2. Sensitive but frequent relapses or steroids dependence nephrotic syndrome
3. No severe hormonal side effects and/or low-dose steroids dependent idiopathic nephrotic syndrome in children (defined as two relapses with an average dose < 0.5mg/kg/day or equivalent alternate-day dose)
4. Normal renal function: eGFR≥90ml/min/1.73m2;
5. Morning urine protein <1+ or urine protein-creatinine ratio <0.2g/g (<20 mg/mmol) for 3 consecutive days and above when in enroll;
6. Prednisone dose was 1.5-2 mg/kg per day before admission;
7. No use of other immunosuppressants (such as tacrolimus, mortecophenolate, cyclosporin A, cyclophosphamide, levamisole, imidazole ribin, or tripterygium, etc.) within 3 months, and no use of rituximab or beliumab within 6 months.

Exclusion Criteria:

1. Family history of nephrotic syndrome, chronic glomerulonephritis, uremia and other kidney diseases;
2. Patients with congenital or acquired immunodeficiency, or with active tuberculosis, active CMV, EBV, hepatitis B, hepatitis C, HIV infection, deep fungal infection, or other active infections;
3. Recurrent or persistent hypertension;
4. Secondary nephrotic syndrome, such as nephrotic syndrome secondary to systemic lupus erythematosus, diabetes, drug poisoning and infection;
5. Combined with other kidney diseases, such as polycystic kidney, ANCA vasculitis, urinary system malformations, etc.;
6. Patients with hypertension, diabetes, tuberculosis, suppurative or fungal infection, gastric and duodenal ulcer disease and heart failure; Patients with other serious heart, liver and other important organs, blood system, endocrine system and other system lesions;
7. Co-occurrence of other monogenic genetic diseases known to affect the condition of nephrotic syndrome;
8. Patients with serious autoimmune diseases or tumors;
9. Use of other immunosuppressants (such as tacrolimus, mortecophenolate, cyclosporin A, cyclophosphamide, levamisole, imidazole ribin, or tripterygium, etc.) within 3 months, and no use of rituximab or beliumab within 6 months;
10. Patients who are known to be allergic to ACTH, glucocorticoids, or any of the components of these drugs, and patients with severe hormone-related side effects
11. History of organ transplantation (excluding corneal and hair transplantation);
12. Patients who had participated in other clinical trials within three months prior to enrollment;
13. Any patient whom the investigator determines is not suitable for inclusion in the trial.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival time(day) within 48 weeks | Within 48 weeks after randomization
  Recurrence-free survival time(day) within 48 weeks

SECONDARY OUTCOMES:
Number of relapses during 48 weeks follow up | Within 48 weeks after randomization
  Number of nephrotic syndrome relapses per patient year during the 48 weeks after randomization
The first time to relapse | Within 48 weeks after randomization
  The first time to relapse after patients taking part in this study
Cumulative prednisone dosage (milligrams per kilogram per year) | Within 48 weeks after randomization
  The total dosage of prednisones from the beginning to the end of the trial
Change in renal function of the patients | Within 48 weeks after randomization
  The change for renal function was judged by the changes of serum creatinine and estimated glomerular filtration rate in each follow-up during the study
Change in anthropometry and growth velocity during 48 weeks after randomization | Within 48 weeks after randomization
  Changes in standard deviation scores for weight, height and body mass index during 48 weeks after randomization
Change in serum cholesterol, hemoglobin and blood albumin of the patients | Within 48 weeks after randomization
  The changes of serum cholesterol, hemoglobin and blood albumin in each follow-up during the study
Incidence of infection | Within 48 weeks after randomization
  The incidence of infection during the study
Adverse event | Within 48 weeks after randomization
  The number of harmful reactions and the types of adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: yi Xie, Study Director — Recruiting
Locations (8):
- China (8):
  - Tongji Hospital, Wuhan, Hubei
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - Kunming Children's Hospital, Kunming, Yunnan
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Women & Children's Hospital, Ningbo, Zhejiang
  - Yuying Childrens Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Children's Hospital affiliated to Capital Institute of Pediatrics, Beijing
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang CS, Greenbaum LA. Nephrotic Syndrome. Pediatr Clin North Am. 2019 Feb;66(1):73-85. doi: 10.1016/j.pcl.2018.08.006. PMID 30454752
- [Background] Wong W. Idiopathic nephrotic syndrome in New Zealand children, demographic, clinical features, initial management and outcome after twelve-month follow-up: results of a three-year national surveillance study. J Paediatr Child Health. 2007 May;43(5):337-41. doi: 10.1111/j.1440-1754.2007.01077.x. PMID 17489822
- [Background] Chakraborty R, Mehta A, Nair N, Nemer L, Jain R, Joshi H, Raina R. ACTH Treatment for Management of Nephrotic Syndrome: A Systematic Review and Reappraisal. Int J Nephrol. 2020 Jun 4;2020:2597079. doi: 10.1155/2020/2597079. eCollection 2020. PMID 32566293
- [Background] Lieberman KV, Pavlova-Wolf A. Adrenocorticotropic hormone therapy for the treatment of idiopathic nephrotic syndrome in children and young adults: a systematic review of early clinical studies with contemporary relevance. J Nephrol. 2017 Feb;30(1):35-44. doi: 10.1007/s40620-016-0308-3. Epub 2016 Apr 16. PMID 27084801
- [Background] Hladunewich MA, Cattran D, Beck LH, Odutayo A, Sethi S, Ayalon R, Leung N, Reich H, Fervenza FC. A pilot study to determine the dose and effectiveness of adrenocorticotrophic hormone (H.P. Acthar(R) Gel) in nephrotic syndrome due to idiopathic membranous nephropathy. Nephrol Dial Transplant. 2014 Aug;29(8):1570-7. doi: 10.1093/ndt/gfu069. Epub 2014 Apr 8. PMID 24714414
- [Background] Hogan J, Bomback AS, Mehta K, Canetta PA, Rao MK, Appel GB, Radhakrishnan J, Lafayette RA. Treatment of idiopathic FSGS with adrenocorticotropic hormone gel. Clin J Am Soc Nephrol. 2013 Dec;8(12):2072-81. doi: 10.2215/CJN.02840313. Epub 2013 Sep 5. PMID 24009220
- [Background] Zand L, Canetta P, Lafayette R, Aslam N, Jan N, Sethi S, Fervenza FC. An Open-Label Pilot Study of Adrenocorticotrophic Hormone in the Treatment of IgA Nephropathy at High Risk of Progression. Kidney Int Rep. 2019 Oct 31;5(1):58-65. doi: 10.1016/j.ekir.2019.10.007. eCollection 2020 Jan. PMID 31922061
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526